CLINICAL TRIAL: NCT07108803
Title: European Research Group on Outcomes of Surgical Treatment of Infective Endocarditis (ERGOSTE)
Brief Title: European Research Group on Outcomes of Surgical Treatment of Infective Endocarditis
Acronym: ERGOSTE
Status: Enrolling by invitation | Type: Observational
Sponsor: Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI) (Unknown)
Responsible Party: Principal Investigator, Giuseppe Gatti, Principal Investigator, Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI)
Other Study IDs: 386_2024
Record Dates: First submitted 2025-07-16; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Infective Endocarditis (IE)
Keywords: Infective endocarditis; Cardiac surgery; Outcomes; Risk score; Prediction; In-hospital mortality; Pathogen agents; Statistics; Sepsis; Surgical techniques; Epidemiology
MeSH Terms: conditions — Endocarditis; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The European Research Group on Outcomes of Surgical Treatment of Infective Endocarditis (ERGOSTE) is a nascent large surgical registry that would encompass most relevant aspects of IE in Europe in the contemporary era.

DETAILED DESCRIPTION:
ERGOSTE, Purposes:

* To create a European multicenter retrospective database including a large number of patients undergoing surgical treatment for infective endocarditis (IE).
* To perform epidemiologic analyses of IE-patients and involved pathogens.
* To find independent predictors of early post-operative death.
* To test ALL the scoring systems specifically developed to predict early death after surgery for infective endocarditis.
* To devise a specific risk score for early postoperative death.
* To explore early and late outcomes of these very difficult patients in order to establish optimal indications, techniques and timing of surgery.
* To carry out a number of sub-analyses concerning the demographic parameters and variable clinical presentation of patients, type and severity of cardiac structural involvement, adopted valve prostheses and surgical techniques, and different involved microbiologic agents.
* To lay experiential foundations of a prospective database on the topic.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery due to infective endocarditis

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery due to infective endocarditis
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Early post-operative mortality | Mortality at 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiac Surgery Unit - ASUGI, Trieste, TRIESTE, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR